CLINICAL TRIAL: NCT04939779
Title: A Randomized, Open-label, Single-dose, Two-way Crossover, Phase 1 Trial to Evaluate Bioequivalence of "LCB01-0371(Batch#1650006)" and "LCB01-0371(Batch#3183817R)" in Healthy Adult Subjects
Brief Title: Trial to Evaluate Bioequivalence of LCB01-0371 in Different Batches
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LCB01-0371-18-1-08
Record Dates: First submitted 2021-02-21; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Healthy
MeSH Terms: interventions — delpazolid; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Period 1: LCB01-0371 tablet 400mg (Reference drug, Batch# 1650006) Period 2: LCB01-0371 tablet 400mg (Test drug, Batch# 3183817R)
  Interventions: Drug: LCB01-0371 tablet 400mg (Test drug, Batch# 3183817R); Drug: LCB01-0371 tablet 400mg (Reference drug, Batch# 1650006)
- Group B (Experimental): Period 1: LCB01-0371 tablet 400mg (Test drug, Batch# 3183817R) Period 2: LCB01-0371 tablet 400mg (Reference drug, Batch# 1650006)
  Interventions: Drug: LCB01-0371 tablet 400mg (Test drug, Batch# 3183817R); Drug: LCB01-0371 tablet 400mg (Reference drug, Batch# 1650006)

INTERVENTIONS:
Drug: LCB01-0371 tablet 400mg (Test drug, Batch# 3183817R) — Oral administration
Drug: LCB01-0371 tablet 400mg (Reference drug, Batch# 1650006) — Oral administration

SUMMARY:
The objective of this clinical trial is to evaluate bioequivalence of "LCB01-0371 (Batch# 1650006)" and "LCB01-0371(Batch#3183817R) in healthy adult subject

ELIGIBILITY:
Inclusion Criteria:

1. A person who is a healthy adult aged between 19 and 45 years old with the result of BMI between 18.0 kg/m2 and 28.0 kg/m2
2. A healthy adult whose weight is over 50 kg
3. A person who is deemed suitable for a clinical trial subject in physical examination, vital sign tests, diagnostic examination, and 12-lead ECG by the medical doctor, etc.

Exclusion Criteria:

1. A person who has a clinically significant history of the disease, such as liver, kidney, gastrointestinal disease, respiratory tract disease, muscular-skeletal disease, endocrine disease, nervous system disease, blood ∙ tumor disease, cardiovascular disease, etc.
2. A person who has a history of gastrointestinal diseases or surgery that may affect the absorption of IP, etc.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic evaluation: The observed maximum concentration(Cmax) | 0-12hours
  Pharmacokinetic parameters will be assessed using non-compartmental method
Pharmacokinetic evaluation:Area under the blood concentration-time curve (AUClast) | 0-12hours
  Area under the plasma concentration curve from zero until the last measurable concentration

SECONDARY OUTCOMES:
Pharmacokinetic evaluation: Time to reach Cmax(Tmax) | 0-12hours
  Pharmacokinetic parameters will be assessed using non-compartmental method
Pharmacokinetic evaluation: Elimination half-life(t1/2) | 0-12hours
  Pharmacokinetic parameters will be assessed using non-compartmental method
Pharmacokinetic evaluation: Apparent total body clearance after extravascular administration(CL/F) | 0-12hours
  Pharmacokinetic parameters will be assessed using non-compartmental method
Pharmacokinetic evaluation:Apparent volume of distribution after extravascular administration(Vd/F) | 0-12hours
  Pharmacokinetic parameters will be assessed using non-compartmental method
Pharmacokinetic evaluation:Area under the blood concentration-time curve (AUCinf) | 0-12hours
  Area under the curve from time 0 extrapolated to infinite time

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koh J, Khwarg J, Cho YL, Yu KS, Chung JY. Comparative pharmacokinetics study of two tablet formulations of delpazolid, a novel oxazolidinone class antibiotic. Transl Clin Pharmacol. 2024 Dec;32(4):216-224. doi: 10.12793/tcp.2024.32.e18. Epub 2024 Dec 18. PMID 39801777